CLINICAL TRIAL: NCT04685135
Title: A Randomized Phase 3 Study of MRTX849 Versus Docetaxel in Patients With Previously Treated Non-Small Cell Lung Cancer With KRAS G12C Mutation
Brief Title: Phase 3 Study of MRTX849 (Adagrasib) vs Docetaxel in Patients With Advanced Non-Small Cell Lung Cancer With KRAS G12C Mutation
Acronym: KRYSTAL-12
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA239-0013; CA239-0013 (Other: Bristol-Myers Squibb Protocol ID); 849-012 (Other: Mirati Therapeutics Protocol ID)
Expanded Access: NCT05162443 (Approved for marketing)
Record Dates: First submitted 2020-12-21; First posted 2020-12-28 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Non Small Cell Lung Cancer; Advanced Non Small Cell Lung Cancer
Keywords: KRAS G12C; Non-small cell lung cancer; NSCLC; Metastatic Cancer; Docetaxel; Phase 3 Clinical Trial; Adagrasib; KRAS; KRAZATI
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — adagrasib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MRTX849 (Experimental)
  Interventions: Drug: MRTX849
- Docetaxel (Active Comparator)
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: MRTX849 — 21 day cycles
  Other Names: adagrasib; KRAZATI
  Arms: MRTX849
Drug: Docetaxel — 21 day cycles
  Other Names: Taxotere
  Arms: Docetaxel

SUMMARY:
This Phase 3 study will evaluate the efficacy of the investigational agent MRTX849 (adagrasib) versus docetaxel in patients who have been previously treated for metastatic NSCLC with a KRAS G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of NSCLC with KRAS G12C mutation.
* Candidacy to receive treatment with docetaxel.

Crossover Inclusion Criteria:

* Evidence of RECIST 1.1 defined disease progression on docetaxel per BICR
* ECOG performance status 0-2

Exclusion Criteria:

* Prior treatment with an agent targeting KRAS G12C (e.g., AMG 510, Sotorasib).
* Active brain metastases.

Crossover Exclusion Criteria:

* Receipt of any other systemic anti-cancer therapy after last administration of docetaxel on the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2026-07-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (343):
- United States (112):
  - Local Institution - 012-898, Cerritos, California
  - City of Hope - Duarte (Main Campus), Duarte, California
  - Local Institution - 012-898 D, Glendale, California
  - Local Institution - 012-910-A, Huntington Beach, California
  - Local Institution - 012-910-C, Irvine, California
  - City Of Hope, Long Beach, California
  - Local Institution - 012-910-F, Long Beach, California
  - Local Institution - 012-910-D, Newport Beach, California
  - Local Institution - 012-898 C, Santa Ana, California
  - Providence Medical Group - Santa Rosa, Santa Rosa, California
  - Local Institution - 012-910-E, Torrance, California
  - Local Institution - 012-951-B, Denver, Colorado
  - SCL Health - Saint Joseph Hospital Cancer Center, Lafayette, Colorado
  - Local Institution - 012-872, Lone Tree, Colorado
  - Local Institution - 012-951-A, Wheat Ridge, Colorado
  - Local Institution - 012-562-B, Fleming Island, Florida
  - Holy Cross Health Fort Lauderdale - Holy Cross Hospital, Fort Lauderdale, Florida
  - 21st Century Oncology of Jacksonville - North Lee Street, Jacksonville, Florida
  - Local Institution - 012-562-D, Jacksonville, Florida
  - Local Institution - 012-562-E, Jacksonville, Florida
  - Local Institution - 012-562-A, Jacksonville, Florida
  - Local Institution - 012-562-C, Jacksonville, Florida
  - Local Institution - 012-562-F, Jacksonville, Florida
  - Local Institution - 012-562-G, Jacksonville, Florida
  - Local Institution - 012-562, Jacksonville, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Orlando Health University of Florida Health Cancer Center - Head and Neck Center, Orlando, Florida
  - USOR - Woodlands Medical Specialists, Pensacola, Florida
  - Local Institution - 012-839, Plantation, Florida
  - University Cancer & Blood Center (UCBC) - Athens, Athens, Georgia
  - Local Institution - 012-835 - A, Austell, Georgia
  - Local Institution - 012-835 - B, Carrollton, Georgia
  - Local Institution - 012-835 - C, Cartersville, Georgia
  - Local Institution - 012-835 - D, Douglasville, Georgia
  - Northwest Georgia Oncology Centers Wellstar - Marietta, Marietta, Georgia
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Local Institution - 012-972 C, Harvey, Illinois
  - Local Institution - 012-972 A, New Lenox, Illinois
  - Illinois Cancer Specialists - Niles, Niles, Illinois
  - Local Institution - 012-972 B, Orland Park, Illinois
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Local Institution - 012-569, Indianapolis, Indiana
  - Local Institution - 012-569 - B, Lafayette, Indiana
  - Local Institution - 012-569 - C, Lafayette, Indiana
  - Local Institution - 012-569 - A, Mooresville, Indiana
  - Franciscan Health Munster, Munster, Indiana
  - Local Institution - 012-942-B, Chanute, Kansas
  - Local Institution - 012-942-C, Dodge City, Kansas
  - Local Institution - 012-942-D, El Dorado, Kansas
  - Local Institution - 012-942-E, Independence, Kansas
  - Local Institution - 012-942-F, Kingman, Kansas
  - Local Institution - 012-942-G, Liberal, Kansas
  - Local Institution - 012-942-H, McPherson, Kansas
  - Local Institution - 012-942-I, Newton, Kansas
  - Local Institution - 012-942-J, Parsons, Kansas
  - Local Institution - 012-942-K, Pratt, Kansas
  - Local Institution - 012-942-L, Salina, Kansas
  - Local Institution - 012-942-M, Wellington, Kansas
  - Local Institution - 012-820, Westwood, Kansas
  - Local Institution - 012-942-A, Wichita, Kansas
  - Local Institution - 012-942, Wichita, Kansas
  - Local Institution - 012-942-N, Winfield, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Local Institution - 012-911 A, New Orleans, Louisiana
  - Tulane University, New Orleans, Louisiana
  - Local Institution - 012-954 - A, Kennebunk, Maine
  - New England Cancer Specialists - Scarborough, Scarborough, Maine
  - Local Institution - 012-954 - B, Topsham, Maine
  - Frederick Health, Frederick, Maryland
  - Local Institution - 012-974-B, Novi, Michigan
  - Local Institution - 012-974-C, Novi, Michigan
  - Ascension Providence Cancer Center - Southfield, Southfield, Michigan
  - Local Institution - 012-974-A, Southfield, Michigan
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Local Institution - 012-841 - A, Billings, Montana
  - St. Vincent Healthcare Cancer Centers of Montana, Billings, Montana
  - Sisters of Charity of Leavenworth Health St. Marys, Billings, Montana
  - Astera Cancer Care - East Brunswick, East Brunswick, New Jersey
  - Local Institution - 012-975 - A, Edison, New Jersey
  - Local Institution - 012-975 - B, Monroe, New Jersey
  - Local Institution - 012-975 - C, Somerset, New Jersey
  - Local Institution - 012-975 - D, Somerville, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - SUNY Upstate Medical University, Syracuse, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Kettering Health Cancer Center - Main Campus, Kettering, Ohio
  - Oregon Oncology Specialists, Salem, Oregon
  - Lifespan Cancer Institute - Rhode Island Hospital, Providence, Rhode Island
  - Local Institution - 012-960-A, Providence, Rhode Island
  - Prisma Health Cancer Institute - Faris Road, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Texas Oncology - Dallas Fort Worth (DFW) - Arlington Cancer Center North, Arlington, Texas
  - Texas Oncology - Dallas Fort Worth (DFW) - South Austin, Austin, Texas
  - US Oncology Research (USOR), Irving, Texas
  - Texas Oncology - Sherman, Sherman, Texas
  - Utah Cancer Specialists - UCS Cancer Center, Salt Lake City, Utah
  - Local Institution - 012-976-A, Salt Lake City, Utah
  - Local Institution - 012-976-B, Salt Lake City, Utah
  - Local Institution - 012-976-C, Salt Lake City, Utah
  - Local Institution - 012-976-D, Salt Lake City, Utah
  - Local Institution - 012-976-E, Salt Lake City, Utah
  - Local Institution - 012-976-F, Salt Lake City, Utah
  - Local Institution - 012-976-G, Salt Lake City, Utah
  - Local Institution - 012-976-H, Salt Lake City, Utah
  - Local Institution - 012-976-I, Salt Lake City, Utah
  - Local Institution - 012-814 - B, Arlington, Virginia
  - UVA Health - University Hospital, Charlottesville, Virginia
  - Local Institution - 012-814 - A, Fairfax, Virginia
  - NEXT Virginia, Fairfax, Virginia
  - Local Institution - 012-814 - C, Gainesville, Virginia
  - Local Institution - 012-814 - D, Leesburg, Virginia
- Australia (8):
  - Local Institution - 012-016, Mackay, Queensland
  - Local Institution - 012-005, Bedford Park
  - Local Institution - 012-004, Clayton
  - Townsville University Hospital, Douglas
  - Local Institution - 012-013, St Leonards
  - Local Institution - 012-019, Tweed Heads
  - Cancer Care Wollongong, Wollongong
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Klinikum Klagenfurt Am Worthersee, Klagenfurt
  - Uniklinikum Salzburg, Salzburg
  - Wiener Gesundheitsverbund - Klinik Ottakring, Vienna
- Belgium (8):
  - Universitair Ziekenhuis Brussel, Brussels
  - Local Institution - 012-157, Edegem
  - Local Institution - 012-155, Ghent
  - Local Institution - 012-151, Gilly
  - Local Institution - 012-158, Hasselt
  - Local Institution - 012-152, Roeselare
  - Algemeen Ziekenhuis Glorieux Ronse, Ronse
  - Local Institution - 012-150, Yvoir
- Czechia (4):
  - Local Institution - 012-164, Hořovice
  - Local Institution - 012-162, Olomouc
  - Vseobecna Fakultni Nemocnice v Praze, Prague
  - Fakultni nemocnice Bulovka, Praha 8 - Liben
- France (23):
  - Local Institution - 012-191-A, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Local Institution - 012-191-B, Lyon, Rhone
  - Local Institution - 012-194, Brest
  - Hopital Louis Pradel, Bron
  - Local Institution - 012-193, Caen
  - Local Institution - 012-196, Caen
  - Centre Hospitalier Intercommunal de Creteil, Créteil
  - Local Institution - 012-192, Dijon
  - LHopital Nord-Ouest (HNO) - Villefranche-sur-Saone, Gleizé
  - Hopital Michallon, La Tronche
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire Dupuytren 1, Limoges
  - Institut Paoli-Calmettes, Marseille
  - Hopital Nord de Marseille, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Hopital Emile Muller, Mulhouse
  - Local Institution - 012-685, Nice
  - Centre Hospitalier de Cornouaille - Hopital Laennec, Quimper
  - Institut de Cancerologie de lOuest - Saint-Herblain - Site Rene Gauducheau, Saint-Herblain
  - Hopital Civil, Strasbourg
  - Local Institution - 012-197, Strasbourg
  - Hopital Bretonneau, Tours
  - Gustave Roussy, Villejuif
- Germany (15):
  - Local Institution - 012-219, Bad Berka
  - Universitatsklinikum Bonn, Bonn
  - Klinikum Koln-Merheim, Cologne
  - Local Institution - 012-210, Essen
  - Local Institution - 012-214, Gauting
  - Local Institution - 012-671, Giessen
  - LungenClinic Grosshansdorf, Grohansdorf
  - Local Institution - 012-215, Halle
  - Universitatsklinikum Jena, Jena
  - Klinikum Kassel, Kassel
  - Local Institution - 012-224, Löwenstein
  - Local Institution - 012-216, Lübeck
  - Local Institution - 012-220, München
  - Local Institution - 012-672, Offenbach
  - Pius-Hospital Oldenburg, Oldenburg
- Greece (11):
  - Henry Dunant Hospital Center, Athens, Attica
  - Local Institution - 012-236, Athens
  - University General Hospital of Heraklion (PAGNI), Heraklion
  - Local Institution - 012-235, Larissa
  - "General Oncology Hospital of Kifisias "Agioi Anargyroi"", Nea Kifissia
  - Local Institution - 012-234, Piraeus
  - Metropolitan Hospital, Piraeus
  - BioClinic Thessaloniki, Thessaloniki
  - Local Institution - 012-230, Thessaloniki
  - Local Institution - 012-500, Thessaloniki
  - Anassa General Clinic, Volos
- Hong Kong (3):
  - Humanity & Health Clinical Trial Centre, Central
  - Prince of Wales Hospital - Hong Kong, Hong Kong
  - Hong Kong United Oncology Centre, Kowloon
- Hungary (7):
  - Local Institution - 012-242, Budapest
  - Local Institution - 012-244, Budapest
  - Local Institution - 012-241, Budapest
  - Local Institution - 012-243, Gyöngyös
  - Local Institution - 012-763, Gyula
  - Local Institution - 012-759, Székesfehérvár
  - Reformatus Pulmonologiai Centrum, Törökbálint
- Ireland (6):
  - The Meath Foundation, Tallaght, Dublin
  - St. Vincents University Hospital, Dublin
  - Beaumont Hospital - Dublin, Dublin
  - St. Jamess Hospital, Dublin
  - University Hospital Galway, Galway
  - University Hospital Limerick, Limerick
- Italy (25):
  - Local Institution - 012-276, Alessandria
  - Local Institution - 012-292, Avellino
  - Local Institution - 012-274, Aviano
  - Local Institution - 012-275, Bari
  - Local Institution - 012-765, Brescia
  - Local Institution - 012-286, Candiolo
  - Local Institution - 012-284, Catania
  - Local Institution - 012-282, Catania
  - Local Institution - 012-762, Florence
  - Local Institution - 012-273, Genova
  - Local Institution - 012-285, Genova
  - Local Institution - 012-279, Lecce
  - "Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - IRST", Meldola
  - Local Institution - 012-296, Milan
  - Local Institution - 012-278, Milan
  - Local Institution - 012-283, Milan
  - Local Institution - 012-271, Napoli
  - Local Institution - 012-277, Napoli
  - Local Institution - 012-770, Novara
  - Local Institution - 012-272, Parma
  - Local Institution - 012-281, Perugia
  - Local Institution - 012-766, Pesaro
  - Local Institution - 012-767, Ravenna
  - Local Institution - 012-295, Roma
  - Local Institution - 012-758, Verona
- Netherlands (7):
  - Local Institution - 012-306, Amsterdam
  - Amphia Ziekenhuis - Breda Molengracht, Breda
  - Local Institution - 012-300, Maastricht
  - Local Institution - 012-630, Nijmegen
  - Local Institution - 012-308, The Hague
  - Local Institution - 012-307, Utrecht
  - Universitair Medisch Centrum Utrecht, Utrecht
- Poland (9):
  - Instytut MSF, Lodz
  - Local Institution - 012-321, Lublin
  - Local Institution - 012-760, Lublin
  - Local Institution - 012-325, Otwock
  - Local Institution - 012-320, Rzeszów
  - Local Institution - 012-324, Skorzewo
  - Wojewodzki Szpital Zespolony im. L. Rydygiera w Toruniu, Torun
  - Local Institution - 012-322, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- Portugal (16):
  - Unidade Local de Saude de Almada-Seixal, E. P. E (Hospital Garcia de Orta), Almada
  - Unidade Local de Saude de Braga, E. P. E (Hospital de Braga), Braga
  - Local Institution - 012-330, Coimbra
  - Local Institution - 012-645, Coimbra
  - Local Institution - 012-333, Guimarães
  - Local Institution - 012-642, Lisbon
  - Local Institution - 012-338-A, Lisbon
  - The Champalimaud Centre for the Unknown, Lisbon
  - Local Institution - 012-338, Lisbon
  - Unidade Local de Saude de Loures-Odivelas, EPE (Hospital Beatriz Angelo), Loures
  - Hospital CUF Porto, Porto
  - Local Institution - 012-331, Porto
  - Local Institution - 012-339, Porto
  - Unidade Local de Saude de Entre Douro e Vouga, E. P. E, Santa Maria da Feira
  - Unidade Local de Saude da Arrabida, E. P. E (Centro Hospitalar de Setubal), Setúbal
  - Unidade Local de Saude de Gaia/Espinho, E. P. E, Vila Nova de Gaia
- Puerto Rico (3):
  - Puerto Rico Medical Research Center, San Juan
  - FDI Clinical Research (Fundacion de Investigacion de Diego) - San Juan, San Juan
  - PanOncology Trials - Rio Piedras Medical Center, San Juan
- Romania (12):
  - Spitalul Jude�ean de Urgen�a dr. Constantin Opri� Baia Mare, Baia Mare
  - SC Policlinica de Diagnostic Rapid SA, Brasov
  - Centrul Oncologic Sanador, Bucharest
  - Local Institution - 012-342, Bucharest
  - Local Institution - 012-344, Cluj-Napoca
  - Local Institution - 012-340, Cluj-Napoca
  - Oncolab Craiova, Craiova
  - Local Institution - 012-343, Craiova
  - Local Institution - 012-513, Iași
  - Ovidius Clinical Hospital, Ovidiu
  - Oncocenter - Oncologie Clinica, Timișoara
  - SC OncoMed SRL, Timișoara
- Russia (11):
  - Evimed Oncology Clinic, Chelyabinsk
  - "Budgetary Healthcare Institution of the Udmurt Republic "Republican Clinical Oncological Dispensary n.a. Sergey Grigoryevich Pr, Izhevsk
  - "Regional Budgetary Healthcare Institution "G.E. Ostroverkhov Kursk Oncology Scientific and Clinical Center" of the Healthcare C, Kislino Village
  - VitaMed - Moscow, Moscow
  - University Headache Clinic, Moscow
  - State Budgetary Healthcare Institution of the Nizhny Novgorod Region Clinical Diagnostic Center, Nizhny Novgorod
  - "Limited Liability Company Medical Sanitary Unit "Clinicist-Clinic Pretor"", Novosibirsk
  - "Budgetary Healthcare Institution of Omsk region "Clinical Oncologic Dispensary"", Omsk
  - Local Institution - 012-355, Saint Petersburg
  - "Federal State Budgetary Institution "Influenza Research Institute named after N.N. A.A. Smorodintsev" of the Ministry of Health, Saint Petersburg
  - Local Institution - 012-354, Saint Petersburg
- Singapore (5):
  - Local Institution - 012-093, Singapore
  - Raffles Hospital, Singapore
  - Icon Cancer Centre Farrer Park, Singapore
  - Oncocare Cancer Centre, Singapore
  - Parkway Cancer Centre - Gleneagles Hospital, Singapore
- South Korea (18):
  - Local Institution - 012-111, Busan
  - Local Institution - 012-522, Busan
  - Local Institution - 012-101, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Local Institution - 012-110, Daegu
  - Local Institution - 012-523, Daegu
  - Local Institution - 012-100, Hwasun-gun
  - Local Institution - 012-103, Incheon
  - Local Institution - 012-102, Junggu
  - Local Institution - 012-520, Seongnam-si
  - Local Institution - 012-112, Seongnam-si
  - Korea University Anam Hospital, Seoul
  - Local Institution - 012-118, Seoul
  - Local Institution - 012-106, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea - Seoul St. Marys Hospital, Seoul
  - Catholic University of Korea St. Vincents Hospital, Suwon
  - Local Institution - 012-107, Suwon
- Spain (29):
  - Clinica Universidad de Navarra - Pamplona, Pamplona, Navarre
  - Local Institution - 012-613, A Coruña
  - Local Institution - 012-769, Alicante
  - Hospital Germans Trias i Pujol, Badalona
  - Local Institution - 012-776, Barakaldo
  - Hospital del Mar - Parc de Salut Mar, Barcelona
  - Local Institution - 012-614, Barcelona
  - Local Institution - 012-612, Barcelona
  - Local Institution - 012-600, Barcelona
  - Local Institution - 012-621, Córdoba
  - Local Institution - 012-764, Girona
  - Local Institution - 012-616, Granada
  - Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas de Gran Canaria
  - Hospital de Leon, León
  - Local Institution - 012-615, Lugo
  - Local Institution - 012-607, Madrid
  - Clinica Universidad de Navarra - Madrid, Madrid
  - Local Institution - 012-606, Madrid
  - Local Institution - 012-601, Madrid
  - Local Institution - 012-609, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Local Institution - 012-626, Majadahonda
  - Local Institution - 012-608, Málaga
  - Local Institution - 012-602, Palma de Mallorca
  - Local Institution - 012-604, Santander
  - Local Institution - 012-629, Seville
  - Consorci Hospital General Universitari de Valencia, Valencia
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Local Institution - 012-603, Zaragoza
- Switzerland (3):
  - Universitatsspital Basel, Basel
  - Spital Simmental-Thun-Saanenland, Thun
  - Kantonsspital Winterthur, Winterthur
- United Kingdom (5):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - NHS Lothian, Edinburgh
  - NHS Greater Glasgow and Clyde, Glasgow
  - University Hospitals of Leicester NHS Trust, Leicester
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barlesi F, Yao W, Duruisseaux M, Doucet L, Martinez AA, Gregorc V, Juan-Vidal O, Lu S, De Bondt C, de Marinis F, Linardou H, Kim YC, Jotte R, Felip E, Lo Russo G, Reck M, Michenzie MF, Yang W, Meade JN, Korytowsky B, Mok TSK; KRYSTAL-12 Investigators. Adagrasib versus docetaxel in KRASG12C-mutated non-small-cell lung cancer (KRYSTAL-12): a randomised, open-label, phase 3 trial. Lancet. 2025 Aug 9;406(10503):615-626. doi: 10.1016/S0140-6736(25)00866-9. PMID 40783289
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Adagrasib: Participants with Non Small Cell Lung Cancer (NSCLC) with KRAS G12C mutation and who have received prior therapy with a platinum-based regimen and an immune checkpoint inhibitor were administered in 3-week cycle with Adagrasib tablet or capsule orally at a starting dose of 600 mg twice a day (BID).
- Docetaxel: Participants with Non Small Cell Lung Cancer (NSCLC) with KRAS G12C mutation and who have received prior therapy with a platinum-based regimen and an immune checkpoint inhibitor were administered in 3-week cycle with intravenous infusion of Docetaxel at 75 mg/m^2 over 1 hour or according to institutional practices.
Period: Overall Study
Arm/Group | Adagrasib | Docetaxel
Started | 301 | 152
Safety Population (Participants who received at least one dose of study treatment.) | 298 | 140
Cross Over (Eligible participants receiving Docetaxel based on physician switched to treatment with Adagrasib) | 0 | 44 (Patients who crossed over from Docetaxel to Adagrasib are included in the Docetaxel arm only.)
Completed | 163 | 83
Not Completed | 138 | 69
Not completed — Death | 126 | 53
Not completed — Withdrawal by Subject | 12 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adagrasib | Docetaxel | Total
Number analyzed (Participants) | 301 | 152 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.6 (8.66) | 63.9 (7.81) | 63.7 (8.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 42 | 150
  Male | 193 | 110 | 303
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 199 | 111 | 310
  Unknown or Not Reported | 94 | 35 | 129
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 135 | 81 | 216
  Black or African American | 0 | 0 | 0
  Asian | 72 | 37 | 109
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Other | 2 | 1 | 3
  Not Reported | 81 | 30 | 111
  Missing | 11 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Per Blinded Independent Central Review
Description: Progression-free survival (PFS) is defined as the time from randomization to the date of progression or death due to any cause, whichever occurs first. 95% CI was obtained using Brookmeyer and Crowley method. Participants who are not observed to have progressed or died are censored at the date of last evaluable tumor assessment. Disease progression assessed as per RECISIST 1.1 was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization to the date of progression or death due to any cause, whichever occurs first (up to approximately 143 weeks)
Population: Intent-To-Treat Population includes all participants who are randomized into this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Adagrasib | Docetaxel
Number analyzed (Participants) | 301 | 152
months | 5.49 [4.53 to 6.67] | 3.84 [2.73 to 4.73]
Statistical Analysis 1: Comparison: Adagrasib vs Docetaxel; Test type: Superiority; p < 0.0001, Log Rank; HR and CI are from stratified Cox proportional hazard model; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.45 to 0.76]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to the date of death due to any cause.
Time Frame: From randomization till death due to any cause (up to approximately 143 weeks)
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Objective Response Rate (ORR) as Per Blinded Independent Central Review
Description: Objective Response Rate (ORR) is defined as the percent of participants documented to have a confirmed complete response (CR) or partial response (PR). CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis < 10 mm). All target lesions must be assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter is used in the sum for target nodes, while the longest diameter is used in the sum for all other target lesions. All target lesions must be assessed. Disease progression was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: From randomization till death or till disease progression or initiation of follow-up anti-cancer therapy or withdrawal of consent prior to minimum efficacy follow-up (up to 143 weeks)
Population: Intent-To-Treat Population includes all participants who are randomized into this study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adagrasib | Docetaxel
Number analyzed (Participants) | 301 | 152
percentage of participants | 31.9 [26.7 to 37.5] | 9.2 [5.1 to 15.0]
Statistical Analysis 1: Comparison: Adagrasib vs Docetaxel; Test type: Superiority; p < 0.0001, Cochran Mantel Haenszel chi-square test; Odds Ratio (OR) = 4.68, 95% CI 2-sided [2.56 to 8.56]

4. Secondary Outcome: Duration of Response (DOR) as Per Blinded Independent Central Review
Description: Duration of Response (DOR) in months is defined as the time from date of the first documentation of objective response (CR or PR) to the first documentation of PD or to death due to any cause in the absence of documented PD. CR was defined as complete disappearance of all target lesions with the exception of nodal disease. All target nodes must decrease to normal size (short axis < 10 mm). All target lesions must be assessed. PR was defined as greater than or equal to 30% decrease under baseline of the sum of diameters of all target measurable lesions. The short diameter is used in the sum for target nodes, while the longest diameter is used in the sum for all other target lesions. All target lesions must be assessed. Disease progression was defined as 20% increase in the sum of diameters of target measurable lesions above the smallest sum observed (over baseline if no decrease in the sum is observed during therapy) with a minimum absolute increase of 5 mm.
Time Frame: First documentation of objective response (CR or PR) to the first documentation of PD or to death due to any cause (Up to approximately 22 months)
Population: Intent-To-Treat Population with Confirmed CR or PR. Intent-To-Treat Population includes all participants who are randomized into this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Adagrasib | Docetaxel
Number analyzed (Participants) | 96 | 14
months | 8.31 [6.05 to 10.35] | 5.36 [2.86 to 8.54]

5. Secondary Outcome: 1-Year Survival Rate
Time Frame: Up to 49 months
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Treatment Emergent Adverse Events (TEAEs) are those that first occur or increase in severity on or after the first dose and not more than 28 days after the last dose, and prior to the initiation of subsequent systemic anti-cancer therapy. An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first dose of treatment (Day 1) till 28 days after last dose (Up to approximately 110 weeks)
Population: Safety Population included all the participants who received at least one dose of the study drug. Docetaxel arm do not include adverse events after initiation of crossover Adagrasib treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Crossover Adagrasib: Eligible participants receiving Docetaxel earlier in the study switched to Adagrasib based on physician decision. Participants were administered with Adagrasib orally at a starting dose of 600 mg twice a day (BID).
Arm/Group | Adagrasib | Docetaxel | Crossover Adagrasib
Number analyzed (Participants) | 298 | 140 | 44
Participants
  Any TEAE | 298 | 138 | 44
  Any Treatment-Related TEAE | 280 | 121 | 41
  Any Treatment-Emergent SAE | 149 | 50 | 20
  Any Treatment-Related Treatment-Emergent SAE | 62 | 23 | 7
  Any TEAE Leading to Discontinuation of Treatment | 40 | 25 | 2

7. Secondary Outcome: Number of Participants With Maximum CTCAE Grade Laboratory Abnormality in Hematology Parameters
Description: Blood samples were collected to assess hematology parameters. Adverse events are graded on a scale from 0 to 4 based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0, with Grade 0 being normal Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization.
Time Frame: From first dose of treatment (Day 1) till 28 days after last dose (Up to approximately 110 weeks)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Adagrasib | Docetaxel | Crossover Adagrasib
Number analyzed (Participants) | 298 | 140 | 44
Participants
  Anemia Grade 0 | 50 | 16 | 5
  Anemia Grade 1 | 155 | 74 | 26
  Anemia Grade 2 | 74 | 34 | 7
  Anemia Grade 3 | 16 | 8 | 3
  Anemia Grade 4 | 0 | 0 | 0
  Anemia Missing | 3 | 8 | 3
  Lymphocytes count decreased Grade 0 | 61 | 33 | 9
  Lymphocytes count decreased Grade 1 | 66 | 20 | 7
  Lymphocytes count decreased Grade 2 | 71 | 33 | 10
  Lymphocytes count decreased Grade 3 | 52 | 23 | 9
  Lymphocytes count decreased Grade 4 | 8 | 3 | 0
  Lymphocytes count decreased Missing | 40 | 28 | 9
  Neutrophils count decreased Grade 0 | 227 | 61 | 32
  Neutrophils count decreased Grade 1 | 10 | 13 | 0
  Neutrophils count decreased Grade 2 | 8 | 7 | 0
  Neutrophils count decreased Grade 3 | 4 | 10 | 1
  Neutrophils count decreased Grade 4 | 8 | 21 | 2
  Neutrophils count decreased Missing | 41 | 28 | 9
  Platelets count decreased Grade 0 | 208 | 113 | 35
  Platelets count decreased Grade 1 | 74 | 13 | 6
  Platelets count decreased Grade 2 | 8 | 3 | 0
  Platelets count decreased Grade 3 | 1 | 0 | 0
  Platelets count decreased Grade 4 | 3 | 0 | 0
  Platelets count decreased Missing | 4 | 11 | 3
  White blood cell decreased Grade 0 | 235 | 72 | 36
  White blood cell decreased Grade 1 | 36 | 14 | 3
  White blood cell decreased Grade 2 | 16 | 15 | 1
  White blood cell decreased Grade 3 | 7 | 24 | 0
  White blood cell decreased Grade 4 | 0 | 4 | 1
  White blood cell decreased Missing | 4 | 11 | 3

8. Secondary Outcome: Number of Participants With Maximum CTCAE Grade Laboratory Abnormality in Chemistry Parameters
Description: Blood samples were collected to assess chemistry parameters. Adverse events are graded on a scale from 0 to 4 based on Common Terminology Criteria for Adverse Events (CTCAE) v5.0, with Grade 0 being normal Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization.
Time Frame: From first dose of treatment (Day 1) till 28 days after last dose (Up to approximately 110 weeks)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Adagrasib | Docetaxel | Crossover Adagrasib
Number analyzed (Participants) | 298 | 140 | 44
Participants
  Alanine Aminotransferase increased Grade 0 | 118 | 118 | 23
  Alanine Aminotransferase increased Grade 1 | 107 | 12 | 11
  Alanine Aminotransferase increased Grade 2 | 23 | 0 | 4
  Alanine Aminotransferase increased Grade 3 | 34 | 0 | 1
  Alanine Aminotransferase increased Grade 4 | 5 | 0 | 0
  Alanine Aminotransferase increased Missing | 11 | 10 | 5
  Hypoalbuminemia Grade 0 | 118 | 55 | 19
  Hypoalbuminemia Grade 1 | 109 | 51 | 13
  Hypoalbuminemia Grade 2 | 58 | 22 | 7
  Hypoalbuminemia Grade 3 | 1 | 0 | 0
  Hypoalbuminemia Grade 4 | 0 | 0 | 0
  Hypoalbuminemia Missing | 12 | 12 | 5
  Hypercalcemia Grade 0 | 260 | 108 | 35
  Hypercalcemia Grade 1 | 24 | 19 | 3
  Hypercalcemia Grade 2 | 1 | 0 | 0
  Hypercalcemia Grade 3 | 0 | 0 | 0
  Hypercalcemia Grade 4 | 1 | 0 | 0
  Hypercalcemia Missing | 12 | 13 | 6
  Hypocalcemia Grade 0 | 230 | 111 | 25
  Hypocalcemia Grade 1 | 45 | 14 | 11
  Hypocalcemia Grade 2 | 11 | 2 | 2
  Hypocalcemia Grade 3 | 0 | 0 | 0
  Hypocalcemia Grade 4 | 0 | 0 | 0
  Hypocalcemia Missing | 12 | 13 | 6
  Alkaline Phosphatase increased Grade 0 | 165 | 109 | 24
  Alkaline Phosphatase increased Grade 1 | 82 | 19 | 14
  Alkaline Phosphatase increased Grade 2 | 31 | 2 | 1
  Alkaline Phosphatase increased Grade 3 | 8 | 0 | 0
  Alkaline Phosphatase increased Grade 4 | 1 | 0 | 0
  Alkaline Phosphatase increased Missing | 11 | 10 | 5
  Amylase increased Grade 0 | 181 | 107 | 31
  Amylase increased Grade 1 | 65 | 11 | 7
  Amylase increased Grade 2 | 16 | 3 | 1
  Amylase increased Grade 3 | 6 | 0 | 0
  Amylase increased Grade 4 | 0 | 0 | 0
  Amylase increased Missing | 30 | 19 | 5
  Aspartate Aminotransferase increased Grade 0 | 103 | 115 | 25
  Aspartate Aminotransferase increased Grade 1 | 133 | 14 | 13
  Aspartate Aminotransferase increased Grade 2 | 27 | 0 | 1
  Aspartate Aminotransferase increased Grade 3 | 20 | 0 | 0
  Aspartate Aminotransferase increased Grade 4 | 3 | 0 | 0
  Aspartate Aminotransferase increased Missing | 12 | 11 | 5
  Bilirubin increased Grade 0 | 251 | 125 | 37
  Bilirubin increased Grade 1 | 24 | 2 | 1
  Bilirubin increased Grade 2 | 9 | 1 | 1
  Bilirubin increased Grade 3 | 1 | 0 | 0
  Bilirubin increased Grade 4 | 2 | 0 | 0
  Bilirubin increased Missing | 11 | 12 | 5
  Creatinine increased Grade 0 | 99 | 99 | 14
  Creatinine increased Grade 1 | 55 | 17 | 9
  Creatinine increased Grade 2 | 126 | 11 | 15
  Creatinine increased Grade 3 | 6 | 3 | 1
  Creatinine increased Grade 4 | 1 | 0 | 0
  Creatinine increased Missing | 11 | 10 | 5
  Fasted Hypoglycemia Grade 0 | 146 | 64 | 18
  Fasted Hypoglycemia Grade 1 | 15 | 4 | 2
  Fasted Hypoglycemia Grade 2 | 1 | 0 | 1
  Fasted Hypoglycemia Grade 3 | 0 | 0 | 0
  Fasted Hypoglycemia Grade 4 | 2 | 0 | 0
  Fasted Hypoglycemia Missing | 134 | 72 | 23
  Lipase Increased Grade 0 | 177 | 109 | 28
  Lipase Increased Grade 1 | 63 | 9 | 7
  Lipase Increased Grade 2 | 27 | 6 | 2
  Lipase Increased Grade 3 | 13 | 0 | 1
  Lipase Increased Grade 4 | 0 | 0 | 0
  Lipase Increased Missing | 18 | 16 | 6
  Hypermagnesemia Grade 0 | 265 | 122 | 37
  Hypermagnesemia Grade 1 | 19 | 4 | 2
  Hypermagnesemia Grade 2 | 0 | 0 | 0
  Hypermagnesemia Grade 3 | 1 | 1 | 0
  Hypermagnesemia Grade 4 | 0 | 0 | 0
  Hypermagnesemia Missing | 13 | 13 | 5
  Hypomagnesemia Grade 0 | 213 | 99 | 29
  Hypomagnesemia Grade 1 | 67 | 25 | 10
  Hypomagnesemia Grade 2 | 5 | 3 | 0
  Hypomagnesemia Grade 3 | 0 | 0 | 0
  Hypomagnesemia Grade 4 | 0 | 0 | 0
  Hypomagnesemia Missing | 13 | 13 | 5
  Non-Fasted Hypoglycemia Grade 0 | 163 | 66 | 22
  Non-Fasted Hypoglycemia Grade 1 | 9 | 8 | 3
  Non-Fasted Hypoglycemia Grade 2 | 1 | 0 | 0
  Non-Fasted Hypoglycemia Grade 3 | 0 | 0 | 0
  Non-Fasted Hypoglycemia Grade 4 | 3 | 0 | 0
  Non-Fasted Hypoglycemia Missing | 122 | 66 | 19
  Hyperkalemia Grade 0 | 206 | 107 | 28
  Hyperkalemia Grade 1 | 54 | 15 | 8
  Hyperkalemia Grade 2 | 20 | 6 | 3
  Hyperkalemia Grade 3 | 5 | 0 | 0
  Hyperkalemia Grade 4 | 1 | 1 | 0
  Hyperkalemia Missing | 12 | 11 | 5
  Hypokalemia Grade 0 | 237 | 114 | 36
  Hypokalemia Grade 1 | 43 | 11 | 2
  Hypokalemia Grade 2 | 0 | 0 | 0
  Hypokalemia Grade 3 | 6 | 3 | 0
  Hypokalemia Grade 4 | 0 | 1 | 1
  Hypokalemia Missing | 12 | 11 | 5
  Hypernatremia Grade 0 | 272 | 130 | 39
  Hypernatremia Grade 1 | 14 | 0 | 0
  Hypernatremia Grade 2 | 0 | 0 | 0
  Hypernatremia Grade 3 | 1 | 0 | 0
  Hypernatremia Grade 4 | 0 | 0 | 0
  Hypernatremia Missing | 11 | 10 | 5
  Hyponatremia Grade 0 | 135 | 95 | 18
  Hyponatremia Grade 1 | 126 | 32 | 19
  Hyponatremia Grade 2 | 17 | 3 | 1
  Hyponatremia Grade 3 | 7 | 0 | 0
  Hyponatremia Grade 4 | 2 | 0 | 1
  Hyponatremia Missing | 11 | 10 | 5
  Hyperuricemia Grade 0 | 185 | 103 | 22
  Hyperuricemia Grade 1 | 98 | 22 | 17
  Hyperuricemia Grade 2 | 0 | 0 | 0
  Hyperuricemia Grade 3 | 0 | 0 | 0
  Hyperuricemia Grade 4 | 0 | 0 | 0
  Hyperuricemia Missing | 15 | 15 | 5

9. Secondary Outcome: Plasma Concentration of Adagrasib
Description: Blood samples were collected for assessment of plasma concentration of Adagrasib. Data for participants for which the dose was reduced after receiving starting dose of 600 mg BID, based on physician decision is presented in separate arms.
Time Frame: Day 1 of Cycle 1 (Pre-Dose and Peak), Cycle 2 (Pre-Dose and Peak), Cycle 3 (Pre-Dose), Cycle 5 (Pre-Dose), Cycle 7 (Pre-Dose) (Each cycle is of 21 days)
Population: The PK evaluable population is defined as patients who received at least one dose of active study drug and had at least one blood sample collected to assess PK concentrations
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- Adagrasib 200 mg BID: Participants with Non Small Cell Lung Cancer (NSCLC) with KRAS G12C mutation and who have received prior therapy with a platinum-based regimen and an immune checkpoint inhibitor were administered with study treatment in 3-week cycle and were administered 200 mg BID Adagrasib orally.
- Adagrasib 400 mg QD: Participants with Non Small Cell Lung Cancer (NSCLC) with KRAS G12C mutation and who have received prior therapy with a platinum-based regimen and an immune checkpoint inhibitor were administered with study treatment in 3-week cycle and were administered 400 mg QD Adagrasib orally.
- Adagrasib 400 mg BID: Participants with Non Small Cell Lung Cancer (NSCLC) with KRAS G12C mutation and who have received prior therapy with a platinum-based regimen and an immune checkpoint inhibitor were administered with study treatment in 3-week cycle and were administered 400 mg BID Adagrasib orally.
- Adagrasib 600 mg QD: Participants with Non Small Cell Lung Cancer (NSCLC) with KRAS G12C mutation and who have received prior therapy with a platinum-based regimen and an immune checkpoint inhibitor were administered with study treatment in 3-week cycle and were administered 600 mg QD Adagrasib orally.
- Adagrasib 600 mg BID: Participants with Non Small Cell Lung Cancer (NSCLC) with KRAS G12C mutation and who have received prior therapy with a platinum-based regimen and an immune checkpoint inhibitor were administered with study treatment in 3-week cycle and were administered 600 mg BID Adagrasib orally.
Arm/Group | Adagrasib 200 mg BID | Adagrasib 400 mg QD | Adagrasib 400 mg BID | Adagrasib 600 mg QD | Adagrasib 600 mg BID
Number analyzed (Participants) | 1 | 2 | 48 | 15 | 295
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 Pre-Dose: number analyzed (Participants) | 1 | 0 | 2 | 15 | 295
  Cycle 1 Day 1 Pre-Dose | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA |  | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA
  Cycle 1 Day 1 Peak: number analyzed (Participants) | 1 | 0 | 2 | 15 | 280
  Cycle 1 Day 1 Peak | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA |  | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA | 556.963 (63.550) | 518.944 (86.625)
  Cycle 2 Day 1 Pre-Dose: number analyzed (Participants) | 1 | 0 | 12 | 2 | 194
  Cycle 2 Day 1 Pre-Dose | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA |  | 1579.040 (54.432) | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA | 2097.813 (67.912)
  Cycle 2 Day 1 Peak: number analyzed (Participants) | 0 | 2 | 15 | 13 | 175
  Cycle 2 Day 1 Peak |  | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA | 2011.347 (39.333) | 2331.298 (59.515) | 2117.333 (62.744)
  Cycle 3 Day 1 Pre-Dose: number analyzed (Participants) | 0 | 0 | 45 | 1 | 130
  Cycle 3 Day 1 Pre-Dose |  |  | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA | 1865.408 (42.930)
  Cycle 5 Day 1 Pre-Dose: number analyzed (Participants) | 0 | 0 | 48 | 11 | 82
  Cycle 5 Day 1 Pre-Dose |  |  | 1114.046 (39.300) | 917.541 (73.596) | 1459.470 (39.094)
  Cycle 7 Day 1 Pre-Dose: number analyzed (Participants) | 0 | 2 | 35 | 7 | 54
  Cycle 7 Day 1 Pre-Dose |  | NA (NA) — Concentrations that are below the limit of quantification (BLQ) are treated as NA | 1062.114 (33.842) | 863.539 (42.917) | 1548.018 (41.166)

10. Secondary Outcome: Change From Baseline in Lung Cancer Symptom Scale (LCSS) Average Total Score
Description: The Lung Cancer Symptom Scale (LCSS) is a disease measure of quality of life which evaluates six major lung cancer symptoms and their effect on overall distress and symptom severity, impact on day-to-day activities, and overall quality of life. This patient reported outcome (PRO) questionnaire assesses the following 6 symptoms items (appetite loss, fatigue, cough, dyspnea, hemoptysis, pain) and 3 summary global items (symptom distress, activity level, overall quality of life) for patients using visual analogue scales (VAS) (100 mm horizontal line) ranging from 0 (best rating) to 100 (worst rating). The LCSS average total score is sum of items 1 to 9 divided by the total number of items ((sum of items 1 to 9)/9) ranging from 0 to 100 where high score represent worst outcome. Least Square Mean and Confidence Interval are from a repeated measures model on the response variable change from baseline in LCSS average total score.
Time Frame: Baseline (Day 1) and up to End of Treatment (Up to approximately 106 weeks)
Population: Intent-To-Treat Population includes all participants who are randomized into this study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a sclae
Arm/Group | Adagrasib | Docetaxel
Number analyzed (Participants) | 301 | 152
Score on a sclae | -4.0 [-7.9 to -0.2] | 3.9 [-0.2 to 8.0]

11. Secondary Outcome: Change From Baseline in Lung Cancer Symptom Scale (LCSS) Average Symptom Burden Index Score
Description: The Lung Cancer Symptom Scale (LCSS) is a disease measure of quality of life which evaluates six major lung cancer symptoms and their effect on overall distress and symptom severity, impact on day-to-day activities, and overall quality of life. This patient reported outcome (PRO) questionnaire for average symptom burden index score assesses the following six items (Appetite loss, fatigue, cough, shortness of breath, blood in sputum, pain) for patients using visual analogue scales (VAS) (100 mm horizontal line) ranging from 0 (best rating) to 100 (worst rating). The average symptom burden score is average of all the 6 items ranging from 0 to 100 where high score represent worst outcome. Least square mean and CI are from a repeated measures model on the response variable change from baseline in average symptom burden index score.
Time Frame: Baseline (Day 1) and up to End of Treatment (Up to approximately 106 weeks)
Population: Intent-To-Treat Population includes all participants who are randomized into this study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a sclae
Arm/Group | Adagrasib | Docetaxel
Number analyzed (Participants) | 301 | 152
Score on a sclae | -5.8 [-9.0 to -2.5] | 3.2 [-0.4 to 6.7]

12. Secondary Outcome: Change From Baseline in Lung Cancer Symptom Scale (LCSS) 3-Item Global Index Score
Description: The Lung Cancer Symptom Scale (LCSS) is a disease measure of quality of life which evaluates six major lung cancer symptoms and their effect on overall distress and symptom severity, impact on day-to-day activities, and overall quality of life. This patient reported outcome (PRO) questionnaire for average 3-item global index score assesses the following 3 items (Distress/severity of symptoms from lung cancer, impact on normal activities, quality of life) for patients using visual analogue scales (VAS) (100 mm horizontal line) ranging from 0 (best rating) to 100 (worst rating). The 3 item global index score is average of all the 3 items ranging from 0 to 100 where high score represent worst outcome. LS mean and CI are from a repeated measures model on the response variable change from baseline in 3-item global index score.
Time Frame: Baseline (Day 1) and up to End of Treatment (Up to approximately 106 weeks)
Population: Intent-To-Treat Population includes all participants who are randomized into this study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a sclae
Arm/Group | Adagrasib | Docetaxel
Number analyzed (Participants) | 301 | 152
Score on a sclae | -3.0 [-20.3 to 14.3] | 15.9 [-2.6 to 34.3]

13. Secondary Outcome: Change From Baseline at End of Treatment in European Quality of Life Five Dimensions Questionnaire (EQ-5D-5L) Visual Analogue Scale Score
Description: The Visual Analogue Score (VAS) is a component of the EQ-5D-5L and assesses the patient's self-rated health using a vertical visual analogue scale where numbered 0 (the worst health you can image) to 100 (the best health you can imageine). The smallest change considered clinically meaningful, is defined as a score difference of 7 points.
Time Frame: Baseline (Day 1) and up to End of Treatment (Up to approximately 106 weeks)
Population: Intent-To-Treat Population includes all participants who are randomized into this study. LS mean and CI are from a repeated measures model on the response variable change from baseline in visual analogue scale.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Adagrasib | Docetaxel
Number analyzed (Participants) | 301 | 152
Score on a scale | 0.1 [-4.4 to 4.5] | -3.7 [-8.5 to 1.1]

14. Secondary Outcome: Change From Baseline at End of Treatment in European Quality of Life Five Dimensions Questionnaire (EQ-5D-5L) Health Utility Index Score
Description: The European Quality of Life 5D-5L Scale (EQ-5D-5L) assesses general health-related quality of life. Health is defined in 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses are coded so that a '1' indicates no problem, and '5' indicates the most serious problem. The responses for the 5 dimensions are combined in a 5-digit number. The EQ-5D-5L health utility index (HUI) is assessed using the Crosswalk algorithm for France based on the individual responses to the 5 EQ-5D-5L domains ranging from -0.594 to 1.000. The smallest change considered clinically meaningful, is defined as a score difference of 0.08 points. Least square mean and CI are from a repeated measures model on the response variable change from baseline in health utility index.
Time Frame: Baseline (Day 1) and up to End of Treatment (Up to approximately 106 weeks)
Population: Intent-To-Treat Population includes all participants who are randomized into this study.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Adagrasib | Docetaxel
Number analyzed (Participants) | 301 | 152
Score on a scale | -0.0350 [-0.0977 to 0.0277] | -0.0914 [-0.1572 to -0.0256]

ADVERSE EVENTS:
Time Frame: All cause mortality and non serious adverse events were reported from first first dose of treatment (Day 1) till 28 days after last dose (Up to approximately 110 weeks). Serious adverse events were collected from date of signing of informed consent form till 28 days after last dose (Up to approximately 111 weeks).
Description: The number at risk for All-Cause mortality represents all randomized participants. The number at risk for serious adverse events and other (Not Including Serious) adverse events represents all participants that received at least 1 dose of study medication.
Arm/Group | Adagrasib | Docetaxel | Crossover Adagrasib
All-Cause Mortality (participants affected / at risk) | 126/301 | 53/152 | 15/44
Serious Adverse Events (participants affected / at risk) | 149/298 | 50/140 | 20/44
Other Adverse Events (participants affected / at risk) | 292/298 | 129/140 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adagrasib (N=298) | Docetaxel (N=140) | Crossover Adagrasib (N=44)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Dyschromatopsia (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Retinopathy (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 2
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 9 | 2 | 1
Asthenia (General disorders) | 1 | 1 | 1
Death (General disorders) | 5 | 0 | 0
Fatigue (General disorders) | 4 | 0 | 0
General physical health deterioration (General disorders) | 6 | 1 | 1
Hyperthermia (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 7 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic cytolysis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic ischaemia (Hepatobiliary disorders) | 1 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0
COVID-19 (Infections and infestations) | 4 | 3 | 0
COVID-19 pneumonia (Infections and infestations) | 3 | 2 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Myelitis (Infections and infestations) | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 11 | 7 | 6
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 4 | 2 | 1
Septic shock (Infections and infestations) | 2 | 0 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0
Viral pericarditis (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 0 | 0
Amylase increased (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 0 | 0
Bilirubin conjugated increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood bilirubin unconjugated increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0
Platelet count decreased (Investigations) | 2 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 1
Weight decreased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 5 | 5
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 1 | 1
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Mental disorder (Psychiatric disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 0 | 0
Glomerulonephritis membranoproliferative (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adagrasib (N=298) | Docetaxel (N=140) | Crossover Adagrasib (N=44)
Anaemia (Blood and lymphatic system disorders) | 91 | 48 | 11
Lymphopenia (Blood and lymphatic system disorders) | 10 | 1 | 4
Neutropenia (Blood and lymphatic system disorders) | 8 | 16 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 24 | 5 | 3
Abdominal pain upper (Gastrointestinal disorders) | 30 | 4 | 3
Constipation (Gastrointestinal disorders) | 49 | 19 | 5
Diarrhoea (Gastrointestinal disorders) | 169 | 42 | 29
Nausea (Gastrointestinal disorders) | 114 | 31 | 15
Stomatitis (Gastrointestinal disorders) | 16 | 13 | 1
Vomiting (Gastrointestinal disorders) | 121 | 12 | 16
Asthenia (General disorders) | 81 | 46 | 9
Fatigue (General disorders) | 68 | 27 | 2
Non-cardiac chest pain (General disorders) | 16 | 6 | 3
Oedema peripheral (General disorders) | 40 | 16 | 7
Pyrexia (General disorders) | 46 | 12 | 5
COVID-19 (Infections and infestations) | 25 | 11 | 2
Pneumonia (Infections and infestations) | 20 | 8 | 4
Urinary tract infection (Infections and infestations) | 9 | 4 | 3
Alanine aminotransferase increased (Investigations) | 99 | 4 | 4
Amylase increased (Investigations) | 30 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 99 | 2 | 5
Blood alkaline phosphatase increased (Investigations) | 49 | 4 | 5
Blood creatine phosphokinase increased (Investigations) | 19 | 0 | 2
Blood creatinine increased (Investigations) | 82 | 4 | 14
Electrocardiogram QT prolonged (Investigations) | 19 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 44 | 6 | 2
Lipase increased (Investigations) | 40 | 3 | 4
Lymphocyte count decreased (Investigations) | 17 | 7 | 4
Neutrophil count decreased (Investigations) | 10 | 23 | 0
Platelet count decreased (Investigations) | 24 | 5 | 1
Weight decreased (Investigations) | 43 | 8 | 2
White blood cell count decreased (Investigations) | 13 | 15 | 0
Decreased appetite (Metabolism and nutrition disorders) | 94 | 34 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 11 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 15 | 3 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 2 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 39 | 9 | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 15 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 22 | 10 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 7 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 32 | 6 | 5
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 11 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 8 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 9 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 22 | 7 | 2
Dizziness (Nervous system disorders) | 20 | 4 | 2
Dysgeusia (Nervous system disorders) | 12 | 9 | 0
Headache (Nervous system disorders) | 22 | 6 | 2
Neuropathy peripheral (Nervous system disorders) | 3 | 11 | 0
Insomnia (Psychiatric disorders) | 18 | 8 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 26 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 57 | 23 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 14 | 8 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 35 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 3 | 0
Rash (Skin and subcutaneous tissue disorders) | 29 | 9 | 2
Hypotension (Vascular disorders) | 16 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/35/NCT04685135/Prot_SAP_000.pdf